CLINICAL TRIAL: NCT07383831
Title: Youth Mentor-Led Brief Interpersonal Psychotherapy for Youth Suicide Prevention
Brief Title: Task-Shifting for Youth Suicide Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24.274; K23MH137405 (NIH)
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation; Depressive Symptoms; Adolescent Mental Health
MeSH Terms: conditions — Suicidal Ideation; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted IPT-A Delivered by Youth Mentors (Experimental): Participants in this arm will receive 6 weekly sessions of an adapted, brief Interpersonal Psychotherapy for Adolescents (IPT-A) delivered by trained youth mentors (n=5) at the partnering youth community centers. The intervention focuses on improving interpersonal functioning, communication skills, and supportive relationships to reduce depressive symptoms, low belongingness, and perceived burdensomeness.
  Interventions: Behavioral: Adapted Brief Interpersonal Psychotherapy for Adolescents (IPT-A LAZOS)
- Usual Community Center Services (Active Comparator): Participants in this arm will continue to receive the standard youth programming and services offered at the participating community centers. This is an individual session focused on active listening.
  Interventions: Other: Usual Community Center Services

INTERVENTIONS:
Behavioral: Adapted Brief Interpersonal Psychotherapy for Adolescents (IPT-A LAZOS) — Adolescents in this intervention will receive 6 weekly sessions of an adaptation of Interpersonal Psychotherapy for Adolescents (IPT-A) delivered by trained youth mentors in youth community centers. The adaptation used a community-participatory research approach to culturally and contextually meet the needs of immigrant-origin inner-city adolescents. The adapted intervention keeps core elements (education, affect identification, and interpersonal skills) and bolsters these skills to target belongingness and burdensomeness, which are factors associated with suicide ideation. Sessions follow a structured, manualized approach. The goal is to reduce depressive symptoms, increase sense of belongingness, and decrease perceived burdensomeness among adolescents with subthreshold depression (score between 4-9 in the PHQ-A).
  Other Names: IPT-A
  Arms: Adapted IPT-A Delivered by Youth Mentors
Other: Usual Community Center Services — Participants in this arm will continue to receive the standard youth programs and services offered by the youth community centers, including mentoring, academic support, and recreational activities. They will not receive BIPT-A.
  Other Names: Usual Care; Standard Youth Programming
  Arms: Usual Community Center Services

SUMMARY:
The goal of this randomized clinical trial is to examine the feasibility, acceptability, and mechanisms of change of a brief adaptation of Interpersonal Psychotherapy for Adolescents (IPT-A), adapted and task-shifted to lay providers (mentors, youth trusted adults) in youth community centers (YCCs) as an upstream approach to suicide.

It focuses on Hispanic adolescents ages 12-17 enrolled in these YCCs. The pragmatic clinical trial will evaluate the acceptability and feasibility of adapted IPT-A delivered by mentors in YCCs and whether adapted IPT-A impacts mechanisms of change (depression symptoms, belongingness, and feeling like a burden to others).

The main questions it aims to answer are:

* Is adpated IPT-A, when delivered by trained youth mentors, feasible and acceptable in youth community centers?
* Does adapted IPT-A target key risk factors (e.g., depressive symptoms, low belongingness, and perceived burdensomeness) associated with suicide ideation? Researchers will compare adolescents randomized to adapted IPT-A (6 sessions) delivered by a trained youth mentor with those receiving usual services at the community center (one individual session focused on active listening).

Participants will:

* Be screened for subthreshold depression using the PHQ-9 adolescent version. Adolescents will be included if they score between 4 and 9 (mild depression). Adolescents with a PHQ-9 score of 10 or higher will not be eligible and will be referred to a licensed mental health provider for appropriate care.
* Be randomized to adapted IPT-A or usual care.
* Youth in the intervention arm will participate in 6 weekly adapted IPT-A sessions with a trained youth mentor focused on education, affect identification, and interpersonal skills.

ELIGIBILITY:
Inclusion Criteria:

1. Parent consent
2. Adolescent consent
3. Enrolled in youth community centers
4. Self-identified as Hispanic or Latine
5. Between 12 and 17 years old.
6. Scoring threshold for depression (4-9) as indicated in the PHQ-A.
7. No current report of suicide ideation with plan or self-harming behaviors

Exclusion Criteria:

1. Not consented to participate in the study
2. Scoring 10 or higher in the PHQ-A, indicating depressive disorder
3. Active suicide ideation (i.e., having thoughts of killing oneself, thinking about how in the past month).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Up to 7 weeks.
  Feasibility of Intervention Measure (FIM) is a self-report 4-item survey (Weiner et al., 2017), which will be used to assess whether the intervention can be successfully carried out (feasible).
Acceptability of the intervention | Up to 7 weeks
  The Acceptability and Appropriateness of Intervention Measure (AIM) assesses whether the intervention is satisfactory (acceptability) and relevant (appropriateness) using 8 items (4 for acceptability, 4 for appropriateness; self-report; Weiner et al., 2017).

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by PHQ-A | Up to 7 weeks.
  Depressive symptoms are one of the study's mechanisms of change associated with passive suicide ideation.
  Using the Patient Health Questionnaire-9 Adolescent (PHQ-A), a 9-item self-report scale, we will assess whether symptoms move in the right direction post-intervention. PHQ-A has been validated with the adolescent and Hispanic populations.
Change in interpersonal factors associated with passive suicide ideation. | Up to 7 weeks.
  Thwarted Belongingness and Perceived Burdensomeness are two factors associated with passive suicide ideation. Based on our study's conceptual framework, these two factors are mechanisms of change targeted by IPT-A LAZOS.
  The Interpersonal Needs Assessment (INQ-15) measures the extent to which individuals believe they belong (i.e., thwarted belongingness; TB) or perceive themselves as a burden to others (i.e., perceived burdensomeness; PB). The INQ-15 showed good internal consistency for TB (0.88) and PB (0.78) among Spanish adolescents aged 12-19 (Perez Rodriguez et al., 2022). We will use this scale to assess whether TB and PB move in the right direction.

OTHER OUTCOMES:
Change in anxiety symptoms | Up to 7 weeks.
  Anxiety often co-occurs with depressive symptoms among adolescents. Thus, we will examine anxiety symptoms. We will use the Generalized Anxiety Disorder (GAD-7), a 7-item self-report scale, to assess anxiety.
Change in experiences with discrimination | Up to 7 weeks.
  Experiences with discrimination have been identified as structural factors associated with suicide ideation among minoritized adolescents. We are using the Everyday Experiences Discrimination Scale (EEDS), a 15-item self-report measure of racial and ethnic discrimination. Reliability scores are 0.88 and 0.81 (Shariff-Marco et al., 2011). We are incorporating this scale based on literature suggesting an association between discrimination, depression, and suicide ideation (Polanco-Roman et al. 2021). EEDS has been used with the Spanish-speaking population and is validated in Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Vélez-Grau, PHD, LCSW, Principal Investigator — Boston College; Laura Mufson, PhD, Study Chair — Columbia University; Susan Witte, PhD, Study Chair — Columbia University
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will use the National Institute of Mental Health (NIMH) Data Archive (NDA). NDA is an NIH-funded collaborative resource that contains harmonized human subjects research data. Data submitted to the NDA is stripped of identifiers.
Supporting Information: Analytic Code
Time Frame: Data will be available at the end of the study in 2029.
Access Criteria: Based on the NDA, the qualified scientific community will have access to de-identified data from the study.
URL: https://nda.nih.gov/nda.